CLINICAL TRIAL: NCT01537211
Title: Microprocessor Knee Versus Mechanical Knee: Impact on Functional Outcomes in Dysvascular Transfemoral Amputees
Brief Title: Functional Outcomes in Dysvascular Transfemoral Amputees
Acronym: CLEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Otto Bock Healthcare (Industry)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director, Rehab Technolgoies and Outcomes Lab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00042823
Record Dates: First submitted 2012-02-07; First posted 2012-02-23 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Transfemoral Amputation; Unilateral Traumatic Amputation of Leg at or Above Knee
Keywords: Dysvascular; amputation; above knee; ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microprocessor knee then Mechanical knee (Experimental)
  Interventions: Device: C leg compared to subject's mechanical leg (Otto Bock)
- Mechanical Knee then Microprocessor knee (Experimental)
  Interventions: Device: C leg compared to subject's mechanical leg (Otto Bock)

INTERVENTIONS:
Device: C leg compared to subject's mechanical leg (Otto Bock) — comparison of different prosthetic knees
  Other Names: Otto Bock
  Arms: Mechanical Knee then Microprocessor knee
Device: C leg compared to subject's mechanical leg (Otto Bock) — comparison of different prosthetic knees
  Other Names: Otto Bock
  Arms: Microprocessor knee then Mechanical knee

SUMMARY:
In older adults, poor circulation in the lower extremities leads to serious health complications including limb loss. In addition, individuals with dysvascular disease also suffer from other co-morbidities like diabetes, coronary and cerebrovascular disease. An individual with a transfemoral (TF) amputation is usually fitted with a prosthetic limb to assist with function, including a prosthetic knee and a prosthetic foot. Currently, dysvascular amputees are given a prosthetic knee based on the basic expectation that they will be functionally stable. This consideration does not address higher levels of function like walking at multiple speeds and over uneven ground. Also, dysvascular amputees are not able to counteract their co-morbidities with a more active lifestyle. Walking is less energy efficient; their traditional prostheses may cause early onset of fatigue and induce a fear of falling. Newer microprocessor knees enable patients with transfemoral amputations to walk on different surfaces and at multiple cadences through better control in swing and stance phases of gait. The impact of the functional differences in the prostheses is not clear and requires additional investigation to clarify the choice of the most appropriate functional prosthesis. The purpose of this study is to compare the functional outcomes with the traditional mechanical knee versus the microprocessor knee (C-leg) in transfemoral amputees.

DETAILED DESCRIPTION:
In older adults, poor circulation in the lower extremities or dysvascular disease can lead to serious health complications. In addition, these individuals also suffer from serious co-morbidities like diabetes and coronary or cerebrovascular disease. Circulatory dysfunction or dysvascular disease is the major cause for amputations in the United States (www.amputee-coalition.orf/fact_sheet/amp_stats_cause.html). Increasing sedentary lifestyles have lead to increased rates of diabetes which has significantly contributed to an increased number of amputations in recent years. The risk of amputation in a diabetic individual is 25 times higher than in the non-diabetic population. The level of amputation that is appropriate for an individual depends on the extent of damage to his/her tissues. Common amputations of the lower extremities in the dysvascular population include the transtibial and transfemoral amputations. The individual having a transtibial or below knee amputation, will be fitted with a prosthetic foot to assist with functional ambulation, while a person with a transfemoral amputation will require both a prosthetic foot and knee for ambulatory purposes. Currently dysvascular amputees are given prostheses based on the goal of returning them to a basic level of function focused primarily on stability. They are considered lower functioning walkers and are expected to use a slow and constant walking speed to ambulate around their homes and are not considered traditional community ambulators. Therefore, they are traditionally given standard mechanical knees which are considered safe, as they provide the ability for only simple single speed house-hold tasks. While this criterion does return the patient to function for basic Activities of Daily Living (ADLs) and walking at a single cadence, it does not empower the patient to counteract the previously existing co-morbidities. Dysvascular amputees tend to be less active predisposing them to a more sedentary lifestyle and exacerbating their risk factors. Their prostheses make them energy inefficient and use more energy for ADLs and functional walking. This causes early onset of fatigue, induces anxiety and fear of falling. Further, they are often depressed, lose motivation and curtail their community interaction. This raises the question if dysvascular amputees are further functionally limited by the prostheses traditionally given to them.

More recently, technology has been used to assist with return to function in the amputee population. Microprocessor (MP) controlled knees are among the technological innovations applied to prostheses to not only return amputees to a basic function, but also with a view to return them to their highest possible function. Over the years, clinical use has shown that traditional knees provide the ability to complete ADLs and basic functions like sit - stand. However, activities like negotiating stairs/steps, walking on uneven ground and self-correction during tripping; functions which reintegrate amputees into unlimited community ambulation and social reintegration require prosthetics which advanced functionality. The Otto Bock C-leg is a MP knee that allows the patient a greater level of control in swing and stance phases of gait. This enables the TF amputee to adjust the requirements of gait during dynamic walking like changing the speed of walking, going up and down stairs and inclines, walking on grass and uneven surfaces and crossing an obstacle. The C-leg has been traditionally given to patients who begin post-amputation rehabilitation at a higher level, but are more expensive than traditionally mechanical knees. In the contrary however, a European study that defined health outcomes in terms of quality-adjusted life year (QALY), indicated that the C-leg showed a QALY gain of €3218 per patient, makes it still financial viable keeping it mind its price tag.. The purpose of this study is to compare the traditional mechanical knee to the microprocessor knee (C-leg) in the dysvascular population. The study will specifically evaluate the potential of microprocessor knees to improve the quality of life in dysvascular transfemoral amputees. This includes identifying if the C-leg can increase the activity level to be classified at a higher level by the Medicare classification from K2 (lower level ambulators) to K3 (more proficient ambulators), along with increasing their social interaction in the community.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with dysvascular transfemoral amputations
* 6 months or more post prosthetic fitting
* Homebound or limited community ambulators post amputation
* Ability to walk > 50m in a 2 min walk test

Exclusion Criteria:

* Traumatic, cancer or genetic amputation
* Co-morbidity that completely prevents physical activity
* Significant skin lesions/ulcers on stump that prevent fitting of prosthesis
* Cognitive deficits or visual impairments that would impair their ability to give informed consent or to follow simple instructions during experiment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, 345 E Superior St, Chicago, Illinois, United States

REFERENCES:
- [Background] Theeven P, Hemmen B, Rings F, Meys G, Brink P, Smeets R, Seelen H. Functional added value of microprocessor-controlled knee joints in daily life performance of Medicare Functional Classification Level-2 amputees. J Rehabil Med. 2011 Oct;43(10):906-15. doi: 10.2340/16501977-0861. PMID 21947182
- [Derived] Jayaraman C, Mummidisetty CK, Albert MV, Lipschutz R, Hoppe-Ludwig S, Mathur G, Jayaraman A. Using a microprocessor knee (C-Leg) with appropriate foot transitioned individuals with dysvascular transfemoral amputations to higher performance levels: a longitudinal randomized clinical trial. J Neuroeng Rehabil. 2021 May 25;18(1):88. doi: 10.1186/s12984-021-00879-3. PMID 34034753

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microprocessor Knee Then Mechanical Knee | Mechanical Knee Then Microprocessor Knee
Started | 4 | 6
Completed | 4 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Microprocessor Knee Then Mechanical Knee | Mechanical Knee Then Microprocessor Knee | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.7) | 60.5 (7.5) | 63.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Community Physical Activity as Measured by GPS
Description: The difference in social mobility (as seen by GPS) between the 2 devices will be measured.
Time Frame: baseline, 1 month with mechanical knee, 1 month with microprocessor knee
Measure: Mean (Standard Deviation); unit: Steps per day
Groups:
- Baseline: Baseline data for participants using their own prosthesis
- Mechanical Knee: Data collected from while participants used the mechanical knee
- Microprocessor Knee: Data collected from while participants used the microprocessor knee
Arm/Group | Baseline | Mechanical Knee | Microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 10
Steps per day | 1749 (2072) | 1625 (1150) | 1257 (1164)

2. Secondary Outcome: Change in 6 Minute Walk Test From Baseline
Description: The 6 Minute Walk Test (6MWT) is an endurance test, which measures the distance a subject can walk indoors on a flat, hard surface over a period of 6 minutes, using assistive devices as necessary. The distance covered during the test is measured with a measuring wheel.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: Feet
Groups:
- Baseline: Baseline data collected while participants used their own personal prosthesis
- Post-mechanical Knee: Data collected from after participants used the mechanical knee for six months
- Post-microprocessor Knee: Data collected from after participants used the microprocessor knee for six months
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
Feet | 434.0 (270.3) | 472.2 (348.6) | 476.4 (361.9)

3. Secondary Outcome: Change in 10 Meter Walk Test Gait Speed From Baseline
Description: Measure of self selected walking speed by measuring the time it takes an individual to walk 10 meters. The test is performed using a "flying start," patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
meters per second | 0.483 (0.152) | 0.645 (0.273) | 0.764 (0.282)

4. Secondary Outcome: Change in Amputee Mobility Predictor Score From Baseline
Description: The Amputee Mobility Predictor (AMP) instrument is used to asses the functional mobility through a standardized sequence of mobility tests while using the prosthesis. Individual tasks are scored and combined, resulting in a total assessment, which is scored out of 47. The minimum score is zero and maximum score on this scale is 47. Higher scores indicate better mobility.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
score on a scale | 30 (8) | 34 (6) | 36 (5)

5. Secondary Outcome: Change in Berg Balance Score From Baseline
Description: The Berg balance scale is used to assess balance during functional activities. It is a performance-based tool, scored between 0 and 56 with higher numbers indicating better balance.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
score on a scale | 35 (10) | 39 (14) | 44 (13)

6. Secondary Outcome: Change in Timed Up and Go Test Time From Baseline
Description: The Timed Up and Go (TUG) test is administered to quantify fall risk and functional mobility. TUG is the time taken for the subject to get up from a chair, walk 3 meters, and sit down. The time for the test to be completed is reported in seconds.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
seconds | 29.95 (16.14) | 29.91 (15.61) | 25.32 (14.14)

7. Secondary Outcome: Change in Four Square Step Test Time From Baseline
Description: The four square step test assesses stepping and change of direction. The subject is asked to walk in a sequence across canes arranged to form four squares. The time to complete the sequence is reported in seconds.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
seconds | 17.96 (5.11) | 19.74 (11.72) | 16.79 (11.17)

8. Secondary Outcome: Change in Modified Falls Efficacy Scale From Baseline
Description: The Modified Falls Efficacy Scale is used to determine falls and near-falls. It is a self-reported 14-item questionnaire filled out by the subject. Subjects answer questions about how confident they are in safely completing various tasks on a scale from 0 to 10, with 10 indicating greater confidence. The score below is the average item-score for the assessment.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
score on a scale | 7.58 (1.24) | 8.61 (1.02) | 9.33 (0.69)

9. Secondary Outcome: Change in Community Participation Indicators From Baseline
Description: The Community Participation Indicators questionnaire will be used to determine community and social participation. It is self-reported outcome measure for community participation. Different questions within the questionnaire correspond to two different aspects of community participation: involvement in life situations and control over participation. These two items are reported first in the table below. The minimum score is 0, and the maximum score is 100. Higher values correspond to higher levels of community participation. These two aspects can be further broken down into percentages of productive activities, social activities, and low-frequency activities performed often enough (the remaining reported values). Each of these percentages has a minimum score of zero and a maximum score of 100, with higher percentages indicating greater satisfaction with the frequency to which the activities are performed.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  Involvement in Life Situations | 49.26 (7.23) | 50.16 (6.25) | 55.83 (18.99)
  Control over Participation | 61.68 (10.57) | 65.28 (10.24) | 74.69 (18.67)
  Percent Social Activities Performed Often Enough | 67.19 (28.66) | 68.62 (33.99) | 72.19 (34.59)
  Percent Productive Activities Performed Enough | 62.96 (39.55) | 76.17 (26.18) | 72.96 (32.55)
  Percent Low-Frequency Activities Performed Enough | 57.88 (33.51) | 61.43 (41.40) | 64.79 (35.87)
  Total Percent of Activities Performed Enough | 63.91 (22.51) | 68.74 (27.97) | 69.98 (25.06)

10. Secondary Outcome: Change in Prosthesis Evaluation Questionnaire (PEQ) From Baseline
Description: The Prosthesis Evaluation Questionnaire (PEQ) will be used to determine prosthesis preference. It is a questionnaire filled out by the subject that is sectioned into validated scales related to usage of the given prosthesis. These validated scales are ambulation, appearance, frustration, perceived response, residual limb health, social burden, sounds, utility, and well being. Items included in these scales are scored between a minimum score of 0 and a maximum score of 100. Reported below are the averages of the validated scales. Thus, the average of each scale has a maximum score of 100 and a minimum score of 0, with a larger value indicating a more positive response.
Time Frame: After 3 month acclimation period to device
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post-mechanical Knee | Post-microprocessor Knee
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  Ambulation | 58.64 (18.76) | 58.28 (18.41) | 81.92 (18.74)
  Appearance | 69.80 (19.86) | 68.78 (15.23) | 85.91 (9.32)
  Frustration | 80.8 (21.6) | 64.1 (28.2) | 90.2 (9.2)
  Perceived Response | 83.81 (13.42) | 87.39 (10.73) | 88.86 (13.39)
  Residual Limb Health | 82.8 (15.1) | 79.9 (8.9) | 85.1 (8.8)
  Social Burdern | 70.59 (23.52) | 76.08 (22.73) | 88.72 (15.92)
  Sounds | 74.20 (25.88) | 72.60 (30.49) | 93.50 (6.62)
  Utility | 67.80 (18.59) | 67.02 (17.92) | 83.92 (11.09)
  Well Being | 70.05 (25.63) | 79.00 (18.81) | 85.44 (10.75)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed, before and after every data collection session, through study completion, up to 12 months.
Groups:
- Microprocessor Knee: The arm reflects time during study participation when the participants were wearing the microprocessor knee.
- Mechanical Knee: The arm reflects time during study participation when the participants were wearing the mechanical knee.
Arm/Group | Microprocessor Knee | Mechanical Knee
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT01537211/Prot_SAP_000.pdf